CLINICAL TRIAL: NCT03669081
Title: A Prospective, Double-blind, Randomized Pilot Study Evaluating the Effects of Toradol and Lyrica Verses Placebo for Pain Control After Donor Nephrectomy (TORPEDO)
Brief Title: Study Evaluating the Effects of Toradol and Lyrica for Pain Control After Donor Nephrectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jeffrey Campsen, Associate Professor of Transplant Surgery, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 00094756
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Results first posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-07

CONDITIONS: Pain, Postoperative
Keywords: live kidney donor; donor nephrectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac; Ketorolac Tromethamine; Pregabalin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toradol and Lyrica (Experimental): Over-Encapsulated Pregabalin 75 mg was administered PO 30 minutes prior to operation; Ketorolac 30 mg IV x 1 was administered in the OR, followed by ketorolac 15 mg IV every 6 hours for 7 doses (or until discharge).
  Interventions: Drug: Ketorolac; Drug: Pregabalin
- Placebo and Standard of Care (Placebo Comparator): Identical placebo oral capsule (same size and color) was administered PO 30 minutes prior to operation; Saline placebo IV x 1 was administered in the OR, followed by saline placebo IV every 6 hours for 7 doses. Standard of care practices maintained.
  Interventions: Drug: Placebo oral capsule; Drug: Saline

INTERVENTIONS:
Drug: Ketorolac — Ketorolac was administered intravenously: 30 mg in the operating room, and 15 mg every 6 hours for 7 doses post-operatively.
  Other Names: Toradol
  Arms: Toradol and Lyrica
Drug: Pregabalin — Pregabalin was administered orally: 75 mg 30 minutes prior to operation.
  Other Names: Lyrica
  Arms: Toradol and Lyrica
Drug: Placebo oral capsule — Placebo oral capsule was administered orally 30 minutes prior to operation.
  Arms: Placebo and Standard of Care
Drug: Saline — Saline was administered intravenously: once in the operating room, and every 6 hours for 7 doses post-operatively.
  Arms: Placebo and Standard of Care

SUMMARY:
The investigators will assess how the use of toradol and pregabalin affects return to bowel function and see if there is a difference in length of hospital stay. Narcotic use can affect bowel function so the investigators hypothesize that use of Toradol will decrease delayed bowel function and aid in a patients discharge and reduction of hospital stay.

DETAILED DESCRIPTION:
Perioperative pain management is a significant challenge following surgery. Many pathways contribute to perioperative pain, including nociceptive, inflammatory, and neuropathic sources. Although opioids have long been a mainstay for perioperative analgesia, other non-opioid therapies have been increasingly used as part of a multimodal analgesic regimen to provide improved pain control while minimizing opioid-related side effects

TORADOL (ketorolac tromethamine), is a nonsteroidal anti-inflammatory drug (NSAID), is indicated for the short-term (up to 5 days in adults), management of moderately severe acute pain that requires analgesia at the opioid level.

Anecdotal evidence has shown that the use of Toradol (Ketorolac) is safe in renal surgery patients. The study team aims to further evaluate this in a pilot study specifically in the population of patient who have donated their kidney in live kidney transplants. The study team will assess how the use of toradol affects return to bowel function and see if there is a difference in length of hospital stay. Narcotic use can affect bowel function so the investigators hypothesize that use of Toradol will decrease delayed bowel function and aid in a patients discharge and reduction of hospital stay. The study team will assess differences in visual analog pain scores and total narcotic consumption, whereas secondary endpoints of urine output, serum creatinine and hemoglobin levels to assess for efficacy and safety.

Pregabalin is prescribed for neuropathic pain. In many studies, preoperative administration of pregabalin reduced postoperative morphine consumption and early postoperative pain.

There will be two arms of the study including:

Arm 1 (pure placebo group): Placebo oral preop then Saline placebo IV x 1 in the OR, then saline placebo IV every 6 hours for 7 doses.

Arm 2: Pregabalin 75mg oral preop, then Ketorolac 30 mg IV x 1 in the OR, then ketorolac 15 mg IV every 6 hours for 7 doses.

Toradol and Lyrica will be used consistent with its FDA approval in terms of dosing, route of administration, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients anticipating donating a kidney in a live kidney donor transplant.

Exclusion Criteria:

* Patients not receiving a donor nephrectomy
* Pregnant, lactating, or nursing mothers
* Medical allergies or history that would otherwise be contraindicated for of a non-steroidal anti-inflammatory drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

REFERENCES:
- [Derived] Campsen J, Call T, Allen CM, Presson AP, Martinez E, Rofaiel G, Kim RD. Prospective, double-blind, randomized clinical trial comparing an ERAS pathway with ketorolac and pregabalin versus standard of care plus placebo during live donor nephrectomy for kidney transplant. Am J Transplant. 2019 Jun;19(6):1777-1781. doi: 10.1111/ajt.15242. Epub 2019 Jan 28. PMID 30589514

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Toradol and Lyrica | Placebo and Standard of Care
Started | 34 | 30
Completed | 33 | 29
Not Completed | 1 | 1
Not completed — Data could not be validated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Toradol and Lyrica | Placebo and Standard of Care | Total
Number analyzed (Participants) | 33 | 29 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 27 | 59
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (11) | 45.1 (12.2) | 44.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 17 | 42
  Male | 8 | 12 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Narcotic Use
Description: Cumulative narcotic use was defined by cumulative morphine equivalents over the course of a patient's hospital course. The Washington State Agency Medical Director's Group Opioid dose calculator was used to provide a total morphine dose equivalent (MDE) for each patient while in the hospital.
Time Frame: 82.25 hours
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Toradol and Lyrica | Placebo and Standard of Care
Number analyzed (Participants) | 33 | 29
mg | 27 [13 to 42.3] | 45 [25 to 70.8]
Statistical Analysis 1: Comparison: Toradol and Lyrica vs Placebo and Standard of Care; Test type: Other — The null hypothesis for the test was no difference between groups; p = 0.006, Wilcoxon (Mann-Whitney) — The significance level for this test was 0.05; We used an exact Wilcoxon rank sum test due to the skewed nature of the morphine equivalents data and the small sample sizes in each group

2. Primary Outcome: Length of Hospital Stay
Description: Primary outcomes include length of hospital stay (LOS).
Time Frame: 82.25 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Toradol and Lyrica | Placebo and Standard of Care
Number analyzed (Participants) | 33 | 29
hours | 51.5 [46.5 to 56] | 57.3 [50.6 to 66.3]
Statistical Analysis 1: Comparison: Toradol and Lyrica vs Placebo and Standard of Care; Test type: Other — The null hypothesis was no difference between groups; p = 0.029, Exact Wilcoxon rank sum test

3. Secondary Outcome: Serum Creatinine Levels at One Year Post-operatively
Description: Renal function was evaluated by following serum creatinine levels for up to one year post-operatively.
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Toradol and Lyrica | Placebo and Standard of Care
Number analyzed (Participants) | 33 | 29
mg/dL | 0.6 [0.6 to 0.7] | 0.7 [0.6 to 0.7]
Statistical Analysis 1: Comparison: Toradol and Lyrica vs Placebo and Standard of Care; The safety outcome was used to power our study.To achieve 90% power at a 2.5% significance level for testing that the post-surgery creatinine increase is at most two-fold (where 1.5 fold is expected), or alternatively for the pre-surgery creatinine group to be ≥0.5 times the post-surgery, we need 17 subjects in the toradol group. This calculation was based on a non-inferiority test (one sided t-test) using a coefficient of variation of 0.25 based on preliminary data; Test type: Non-Inferiority — We conducted a 1-sided non-inferiority test using an alpha level of 0.025, for a comparison of the fold change of creatinine levels (pre-operative creatinine/post-operative creatinine) in the Toradol group. Our minimum non-inferiority margin was 0.5, ie the post-operative creatinine level could only increase to at most two times the pre-operative creatinine level; p < 0.0001, Wilcoxon (Mann-Whitney) — This p-value was compared to a significance threshold of 0.025

4. Secondary Outcome: Bleeding Risk
Description: Hematocrit levels were evaluated post-operatively for up to a day post-operatively for signs of blood loss.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percentage of hematocrit
Arm/Group | Toradol and Lyrica | Placebo and Standard of Care
Number analyzed (Participants) | 33 | 29
percentage of hematocrit | 6.3 (2.1) | 4.3 (2.5)
Statistical Analysis 1: Comparison: Toradol and Lyrica vs Placebo and Standard of Care; Test type: Other — The null hypothesis was no difference between groups; p = 0.002, t-test, 2 sided

5. Secondary Outcome: Number of Patients With Urinary Retention
Description: Patients were evaluated post-operatively during hospital stay for instances of urinary retention.
Time Frame: 82.25 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Toradol and Lyrica | Placebo and Standard of Care
Number analyzed (Participants) | 33 | 29
Participants | 1 | 0
Statistical Analysis 1: Comparison: Toradol and Lyrica vs Placebo and Standard of Care; Test type: Other — The null hypothesis was no difference between groups; p > 0.99, Fisher Exact

6. Secondary Outcome: 30 Day Mortality
Description: Primary outcomes include 30 day mortality post-operatively.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Toradol and Lyrica | Placebo and Standard of Care
Number analyzed (Participants) | 33 | 29
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Toradol and Lyrica | Placebo and Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/29
Other Adverse Events (participants affected / at risk) | 0/32 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT03669081/SAP_000.pdf
  • Study Protocol (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT03669081/Prot_001.pdf